CLINICAL TRIAL: NCT05226013
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Tolerance, Pharmacokinetics / Pharmacodynamics (PK / PD) and Immunogenicity of Pegylated Uric Acid Oxidase for Injection in Healthy Adults and Hyperuricemia Volunteers
Brief Title: Tolerance, Pharmacokinetics / Pharmacodynamics (PK / PD) and Immunogenicity of Pegylated Uric Acid Oxidase for Injection in Healthy Adults and Hyperuricemia Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: XZ-PEG-UOX-001
Record Dates: First submitted 2022-01-28; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEGylated Urate Oxidase for Injection (Experimental): PEGylated Urate Oxidase for Injection，specification:5mg，Single dose ascending.Healthy subjects were divided into three dose groups (0.5mg, 1mg, 2mg), and hyperuricemia patients were divided into four dose groups (2mg, 4mg, 8mg, 12 mg), with increasing dose design.Each group will receive the experimental drug in 6 subjects.
  Interventions: Drug: Polyglycol lated urate oxidase for injection
- Placebo (Placebo Comparator): Placebo , specification: 5mg,Single dose. Groups received the placebo in 2 patients per group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyglycol lated urate oxidase for injection — Single dose escalation
  Arms: PEGylated Urate Oxidase for Injection
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study of tolerance, pharmacokinetic / pharmacodynamics (PK / PD) and immunogenicity of single administration of PEG uric oxidase for injection in healthy adults and hyperuricemia volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * Subjects understand well trial purpose, nature, content, process and possible adverse reactions, and voluntarily sign an informed consent form.
  * Serum uric acid level<360 µ mol / L twice on different days.
  * Healthy male or female aged between 18 and 60 years old (including the critical value).
  * The body mass index is in the range of 18-30kg/m2 (including the critical value). The weight of male is not less than 50 kg, and that of female is not less than 45 kg (including the critical value).
  * Subjects who had not any medical history of cardiovascular, digestive, respiratory, nervous, haemal diseases or hepatic/renal impairment.The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: physical examination, 12-lead ECG, vital sign measurements and laboratory safety tests .
  * The subjects have no family planning within 6 months and could select contraceptive method. They have no sperm and egg donation program.
  * Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.
  * The blood pregnancy test of female subjects was negative, the menstrual cycle was regular, and the menstrual bleeding period was 3 ~ 7 days.

Patients with hyperuricemia:

* Patients with hyperuricemia ,male or female aged between 18 and 60 years old (including the critical value).
* Stop uric acid lowering treatment for at least 7 days, and 480≤UA≤540µmol/L twice on different days within 7 days.
* The body mass index is in the range of 18-30kg/m2 (including the critical value). The weight of male is not less than 50 kg, and that of female is not less than 45 kg (including the critical value).
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.
* The blood pregnancy test of female subjects was negative, the menstrual cycle was regular, and the menstrual bleeding period was 3 ~ 7 days.

Exclusion Criteria:

* Healthy volunteers:

  * A history of drug allergy, or allergic allergic disease, or known to be allergic to the test drug or its excipients or the same type of drug;
  * Hepatitis (including hepatitis B and C), positive screening results for AIDS or syphilis;
  * Any history of acute or chronic illness that might affect drug absorption, and/or metabolism;
  * Any history of drug abuse in the past 12 months prior to screening;
  * Any history of alcohol abuse 3 months prior to screening or moderate drinkers (drink more 2 units per day or 14 units per week);
  * Smoking more than 5 cigarettes per day during the 3 months prior to screening;
  * Blood donation, massive blood loss (#400mL) or enrolled in other clinical trials 3 months prior to screening;
  * Any use of other prescription drugs (including contraceptive)#over-the counter drugs, Chinese herbal medicine, health care products and 14 days prior to medication for this study;
  * Any history of postural hypotension, syncope, or amaurosis;
  * 6-glucose phosphate dehydrogenase (G6PD) deficiency;
  * Lactating or pregnant women

Patients with hyperuricemia:

* Using uric acid lowering drugs and unwilling to stop existing drugs.
* Ultrasonic examination of the metatarsal-toe joint suggested the presence of tophi.
* Serum CA72-4 level ≥7.5U / mL.
* History of organic heart disease (symptomatic cardiac insufficiency with grade II-IV).
* Patients with refractory hypertension.
* Patients with malignant tumors (treatment or not).
* Patients with organ transplantation treated with immunosuppressants.
* Any history of drug abuse in the past 12 months prior to screening;
* Any history of alcohol abuse 3 months prior to screening or moderate drinkers (drink more 2 units per day or 14 units per week).
* Smoking more than 5 cigarettes per day during the 3 months prior to screening.
* A history of drug allergy, or allergic allergic disease, or known to be allergic to the test drug or its excipients or the same type of drug.
* Any history of acute or chronic illness that might affect drug absorption, and/or metabolism.
* 6-glucose phosphate dehydrogenase (G6PD) deficiency.
* Once treated with urate oxidase.
* Subjects had an uncorrected dehydration, acidosis, hypotension, renal insufficiency, or were using drugs with nephrotoxicity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 500 days
  Evaluation of Peak Plasma Concentration (Cmax)
Maximum tolerated dose Maximum tolerated dose | 500 days
  Maximum tolerated dose Maximum tolerated dose for a single dose
Area under the plasma concentration versus time curve (AUC)0-t | 500 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t

SECONDARY OUTCOMES:
Occurrence rate of Adverse Events | 500 day
  Adverse events were recorded to evaluate the safety of the studied drugs
Immunogenicity | 500day
  Antidrug antibody detection

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University; Changgui Li, Doctor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Revised Biomedical (Hangzhou) Research Institute Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor.

REFERENCES:
- [Derived] Sun F, Zhang J, Yan Z, Yu Q, Wang P, He Y, Liu M, Huang B, Fang L, Xu Y, Fu Y, Gao X, Li C, Cao Y. Efficacy and safety of PEGylated uricase in healthy adults and patients with hyperuricaemia: A phase I, randomized, double-blind, dose-escalation, placebo-controlled trial. Diabetes Obes Metab. 2025 Sep;27(9):4892-4902. doi: 10.1111/dom.16532. Epub 2025 Jun 25. PMID 40557749
- [Derived] Sun F, Wang C, Xu Y, Lin P, Cao Y, Zhang J, Li X, Jiang X, Fu Y, Cao Y. Randomized, Double-Blind, Placebo-Controlled, Phase I, Dose- Escalation Study to Evaluate the Tolerance, Pharmacokinetics, Pharmacodynamics and Immunogenicity of PEGylated Urate Oxidase for Injection in Healthy Adults and Hyperuricemia Volunteers: Study Protocol. Diabetes Metab Syndr Obes. 2023 Dec 28;16:4263-4268. doi: 10.2147/DMSO.S429114. eCollection 2023. PMID 38164417